CLINICAL TRIAL: NCT00002415
Title: A Phase II, Randomized, Double-Blind, Placebo-Controlled Study of the Safety and Antiviral Activity of the Addition of PMPA Prodrug to Combination Antiretroviral Regimens in Treatment-Experienced HIV-Infected Patients
Brief Title: Safety and Effectiveness of Adding PMPA Prodrug to an Anti-HIV Drug Combination to Treat HIV-Infected Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 283B; GS-98-902
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1999-11

CONDITIONS: HIV Infections
Keywords: Drug Therapy, Combination; Prodrugs; Anti-HIV Agents
MeSH Terms: conditions — HIV Infections | interventions — Tenofovir

INTERVENTIONS:
Drug: Tenofovir disoproxil fumarate

SUMMARY:
The purpose of this study is to see if it is safe and effective to add PMPA Prodrug (a new anti-HIV drug) to an anti-HIV drug combination taken by patients who have taken anti-HIV drugs in the past. Genetic response will be studied.

DETAILED DESCRIPTION:
Prior to study entry patients are stratified according to HIV-1 RNA level, CD4 cell count, and number of antiretroviral drugs. PMPA Prodrug or placebo is added to current antiretroviral regimens, and is administered in one of three dosing regimens. Patients randomized to receive placebo are eligible to receive open-label PMPA Prodrug for the remainder of the 48-week study period after at least 24 weeks post randomization.

ELIGIBILITY:
Inclusion Criteria

You may be eligible for this study if you:

* Are HIV-positive.
* Have an HIV count of 400 - 50,000 copies/ml.
* Are expected to live for at least 1 year.
* Have been taking the same anti-HIV drug combination (made up of no more than 3 anti-HIV drugs) for at least 8 weeks prior to study entry.
* Are at least 18 years old.
* Agree to use effective methods of birth control during the study.

Exclusion Criteria

You will not be eligible for this study if you:

* Have taken medications for certain infections within 15 days prior to study entry.
* Have a history of cancer, except Kaposi's sarcoma (KS) or skin cancer.
* Develop a new AIDS-related condition within 30 days of study entry.
* Have certain serious medical conditions, including severe nausea, vomiting, or other stomach problems that make you unable to take medications by mouth.
* Have received a vaccine within 30 days prior to study entry.
* Have taken certain medications, including those that may affect your kidneys.
* Abuse alcohol or drugs.
* Are pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - Univ of Alabama at Birmingham / 1917 Rsch Cln, Birmingham, Alabama
  - McDowell Clinic, Phoenix, Arizona
  - East Bay AIDS Ctr, Berkeley, California
  - Tower Infectious Disease Med Ctr, Los Angeles, California
  - UCSD Treatment Ctr, San Diego, California
  - San Francisco Veterans Adm Med Cntr, San Francisco, California
  - Harbor UCLA Med Ctr, Torrance, California
  - Univ of Colorado Health Sciences Ctr, Denver, Colorado
  - Hillsborough County Health Dept Special Care Ctr, Tampa, Florida
  - AIDS Research Consortium of Atlanta Inc, Atlanta, Georgia
  - Grady Mem Hosp, Atlanta, Georgia
  - Private Practice / Thacker and Thompson, Atlanta, Georgia
  - Northstar Med Clinic, Chicago, Illinois
  - CRI New England, Brookline, Massachusetts
  - Univ of Minnesota, Minneapolis, Minnesota
  - Beth Israel Med Ctr, New York, New York
  - Cornell Clinical Trials Unit - Chelsea Clinic, New York, New York
  - Univ Hosps of Cleveland, Cleveland, Ohio
  - The Research and Education Group, Portland, Oregon
  - Hershey Med Ctr, Hershey, Pennsylvania
  - Anderson Clinical Research, Pittsburgh, Pennsylvania
  - Roger Williams Med Ctr, Providence, Rhode Island
  - Amelia Ct Clinic, Dallas, Texas
  - Thomas Street Clinic, Houston, Texas

REFERENCES:
- [Background] Miller MD, Margot NA, Schooley R, McGowan I. Baseline and week 48 final phenotypic analysis of HIV-1 from patients adding tenofovir disoproxil fumarate (TDF) therapy to background ART. 8th Conf Retro and Opportun Infect. 2001 Feb 4-8 (abstract no 441)
- [Background] Schooley R, Myers R, Ruane R, Beall G, Lampiris H, McGowan I. A double-blind, placebo-controlled study of tenofovir disoproxil fumarate (TDF) for the treatment of HIV infection. 39th Intersci Conf Antimicrob Agents Chemother. 1999 Sep (abstract no I302I)